CLINICAL TRIAL: NCT03808025
Title: Opioid Use in Shoulder Arthroplasty Patients: A Stratification and Algorithm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1333215
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients who consent to the study will be prospectively randomized to one of two arms: one will receive educational intervention, the other will not. Investigators will be masked to patient intervention when assessing and collecting outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- education (Experimental): The teaching arm would consist of a standardized dialogue the surgeon will complete with the patient in order to familiarize the patient with the risks of over-prescribing opioid medication and set patient expectations regarding the clinic's opioid prescribing pattern protocol, in an effort to minimize the number of opioid pills prescribed or refills required, the amount actually used, and the untoward side effects of opioid use (e.g. respiratory depression, nausea, sedation, restriction from driving, and access to and use by those the medication was not intended).
  Interventions: Behavioral: opioid education
- no education (No Intervention): Standard preoperative care without dedicated teaching regarding opioid use and risks

INTERVENTIONS:
Behavioral: opioid education — see arm/group descriptions
  Arms: education

SUMMARY:
The investigators aim to better understand opioid use in patients undergoing elective shoulder surgery. The investigators will prospectively determine actual postoperative opioid use, while evaluating whether implementation of an educational session with pain contract would help minimize opioid use.

DETAILED DESCRIPTION:
The investigators aim to better understand opioid use in patients undergoing elective shoulder surgery. As part of a multi-part investigation, The investigators intend to prospectively determine actual postoperative opioid use, while evaluating whether implementation of an educational session with pain contract would help minimize opioid use. Through use of a teaching session and pain contract, it is hypothesized opioid use would decrease. The investigators hypothesize the use of a pain contract and thorough discussion regarding proper opioid use and side-effects, will decrease the amount of postoperative opioid use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with capacity to consent
* presenting to UC Davis Medical Center Department of Orthopedic Surgery and planning to undergo elective shoulder surgery

Exclusion Criteria:

* unable to consent
* prisoners
* children
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Opioid use | 6 months after surgery
  Total opioid use

SECONDARY OUTCOMES:
Number of refills | 6 months after surgery
  Necessary refills related to surgical pain

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Szabo, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Department of Orthopaedic Surgery, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-opioid-use-in-shoulder-arthroplasty-patients-139543/